CLINICAL TRIAL: NCT00717184
Title: A Pilot Study of Autologous Ex Vivo Activated NK Cell Infusion in the Treatment of Metastatic Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: NP01/02/06
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Metastatic Nasopharyngeal
MeSH Terms: interventions — Interleukins

INTERVENTIONS:
Drug: Interleukin, NK cells

SUMMARY:
1. To demonstrate the feasibility of leukapheresis and ex vivo activation of autologous NK cells in patients with metastatic NPC
2. To demonstrate the safety of low dose systemic IL-2 in combination with escalating doses of autologous Ex Vivo Activated NK cells in patients with metastatic NPC
3. To assess immune measurements such as quantitation of regulatory T cells, EBV specific T cells, serum cytokine levels, and NK cell function after treatment with IL-2 and autologous Ex Vivo Activated NK cells

DETAILED DESCRIPTION:
We are investigating the use of immune cell therapy in metastatic Nasopharyngeal Cancer (NPC). Recent small studies have shown that EBV specific cytotoxic T cells can be infused into NPC patients with some good clinical effect including tumor responses. We are trying to achieve a similar result using a less complex and less costly approach, with Natural Killer (NK) cells. NK cells are known to recognize tumor and virally infected cells through a variety of mechanisms. Also, NK cells influence the development of antigen-specific T cell responses via reciprocal interactions with dendritic cells and the secretion of IFNγ.

This is a pilot clinical trial to study the feasibility of collecting, manipulating , and infusing autologous enriched NK cells activated by short-term incubation in IL-2. Leukapheresis units will be collected from eligible patients with NPC. NK cells will be selected and activated with IL-2 prior to re-infusion. Patients will receive low dose IL-2 after infusion of activated NK cells. Post infusion monitoring will include peripheral blood T cell subsets, cytokine secretion and serum cytokine levels. The parameters will be correlated to clinical observations. If clinical efficacy is shown, our protocol could represent a simple way of harnessing the immune system of the patient for treatment of this disease. This study will also serve as platform technology development for later trials involving manipulating cell therapy products.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven, metastatic nasopharyngeal carcinoma (NPC) (WHO grade III) and measurable metastatic disease.
* ECOG performance status <2.
* Life expectancy greater than 6 months.
* Patient must have adequate access for leukapheresis (vein or central line)
* Patients must have normal organ and marrow function as defined below:

  1. leukocytes >3,500/μl, absolute neutrophil count >1,500/μl, platelets >100,000/μl.
  2. Organ function tests:
  3. total bilirubin <1.5X normal, AST(SGOT) / ALT(SGPT) <2.5 X of normal or <5X in the case of patients with liver metastases;
  4. creatinine <1.5X normal institutional limits or a calculated creatinine clearance of > 50 mls/min.
* Negative pregnancy test within 4 weeks of enrollment in women of child-bearing age.
* Patients with fertility/child bearing potential must agree to avoid pregnancy.
* Age 18 and older
* Patients must have received at least one prior systemic treatments for "metastatic nasopharyngeal carcinoma".Neoadjuvant chemotherapy or concurrent chemoradiation administered for localized disease does is not considered a line of prior treatment.
* Patient's last dose of systemic chemotherapy must have been given at least 4 weeks prior to the beginning of study treatment. Local radiation therapy will be allowed only if there are other sites of measurable disease.
* Patients must have at least one site of measurable disease. Sites of measurable disease which has been irradiated can be used if greater than 60 days has passed between the completion of radiation treatment and the start of NK cell treatment.

Exclusion Criteria:

* Patients with active infections requiring oral or intravenous antibiotics are not eligible for entry onto the study until resolution of the infection.
* History of HIV infection, chronic active Hepatitis B or C.
* Patients with prior or currently active autoimmune disease requiring management with systemic immunosuppression are not eligible. Asthma or chronic obstructive pulmonary disease that does not require daily systemic corticosteroids is acceptable.
* Enrollment on another experimental treatment within 28 days of starting treatment on this study.
* Systemic steroids within 28 days of starting study treatment.
* Uncontrolled medical problems.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Alvin Seng Cheong Wong, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Farag SS, Caligiuri MA. Human natural killer cell development and biology. Blood Rev. 2006 May;20(3):123-37. doi: 10.1016/j.blre.2005.10.001. Epub 2005 Dec 20. PMID 16364519